CLINICAL TRIAL: NCT00139932
Title: A Double-Blind Randomized, Parallel-Group, Multicenter Clinical Study to Compare the Efficacy and Tolerability of Tiotropium Bromide Alone vs. the Co-Administration of Tiotropium Bromide and Formoterol Fumarate in Subjects With COPD
Brief Title: Tiotropium Bromide Alone vs Tiotropium Bromide and Formoterol Fumarate in Subjects With COPD (Study P04272)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Integrated Therapeutics Group (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04272
Record Dates: First submitted 2005-08-30; First posted 2005-08-31 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: formoterol fumarate

SUMMARY:
This study is being conducted to determine if the co-administration of formoterol fumarate and tiotropium bromide is more effective than the use of tiotropium bromide alone in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinical history of COPD.
* Subjects must be current cigarette smokers or ex-smokers who stopped smoking at least 3 months prior to screening visit (V1). Subjects must have a smoking history of at least 10 pack-years (20 cigarettes per pack). Pack-years are calculated by multiplying the average packs of cigarettes smoked per day times the number of years.
* Subjects on stable inhaled corticosteroids are allowed to be enrolled and to remain on the treatment throughout the study.
* Subjects must be willing to give written informed consent and able to adhere to dose and visit schedules.
* Subjects must agree to inform their usual treating physician of their participation in this study.
* Female subjects of childbearing potential must have a negative urine pregnancy test prior to the randomization of the study
* Nonpregnant women of childbearing potential must be using a medically acceptable, adequate form of birth control.

Exclusion Criteria:

* Subjects have a current or past history of clinically relevant asthma.
* Subjects quit smoking less than 3 months prior to the Screening visit (V1).
* Subjects have required ventilator support for respiratory failure within the last year.
* Subjects have clinically significant lung disease other than COPD, e.g., bronchiectasis, sarcoidosis, pulmonary fibrosis, tuberculosis, etc.
* Subjects have undergone lobectomy, pneumonectomy or lung volume reduction surgery.
* Subjects have had lung cancer diagnosed or treated within the last five years.
* Subjects require nasal continuous positive airway pressure (CPAP) or bi-level positive airway pressure (Bi-PAP).
* Subjects have initiated pulmonary rehabilitation within the past 3 months.
* Subjects use oxygen >= 2 liters per minute for > 2 hours per day.
* Subjects require chronic or prophylactic treatment with antibiotics.
* Subjects have significant renal, hepatic, cardiovascular (including cor pulmonale), metabolic, neurologic, hematologic, gastrointestinal, cerebrovascular or other significant medical illness or disorder which, in the judgment of the Investigator, may interfere with the study or require treatment which may affect the evaluation of efficacy and safety of the study drug.
* Subjects have clinically significant abnormalities on chest x-ray (other than evidence of COPD) at the Screening visit or within the previous year.
* Women are pregnant or breast-feeding.
* Subjects cannot adhere to the concomitant medications restrictions and prohibitions.
* Subjects have used any investigational product within 30 days, or 3 months for any biologic of unknown half-life, prior to the Baseline Visit (V3).
* Subjects are part of the staff or a family member of the staff personnel directly involved with this study.
* Subjects have chronic narrow-angle glaucoma.
* Subjects have symptomatic prostatic hyperplasia or bladder-neck obstruction.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2005-09-01 (Actual); Primary Completion 2006-11-21 (Actual); Study Completion 2006-11-21 (Actual)

PRIMARY OUTCOMES:
effects of tiotropium bromide alone vs.the effect of tiotropium bromide and formoterol fumarate | 12 weeks
  To compare the effects of tiotropium bromide alone vs. the effects of co-administration of tiotropium bromide and formoterol fumarate on the change from baseline of the normalized area under the time curve (AUC) for FEV1 for the 0 hour to 4 hours post-morning dose at the last study visit.

REFERENCES:
- [Result] Tashkin DP, Pearle J, Iezzoni D, Varghese ST. Formoterol and tiotropium compared with tiotropium alone for treatment of COPD. COPD. 2009 Feb;6(1):17-25. doi: 10.1080/15412550902724073. PMID 19229704
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html